CLINICAL TRIAL: NCT06512571
Title: The Characteristics of Cardiovascular Imaging Alterations in Patients with Fabry Cardiomyopathy: a Prospective, Multicenter, Observational Cohort Study
Brief Title: CVI Alterations in FD: a Prospective, Multicenter, Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-ZX084
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease, Cardiac Variant
MeSH Terms: conditions — Fabry Disease, Cardiac Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Fabry disease (FD) is a rare X-linked lysosomal storage disorder caused by α-galactosidase A (GLA) gene mutations leading to reduced or undetectable α galactosidase A (α-Gal A) enzyme activity, resulting in progressive accumulation of globotriaosylceramide (GL3) and its deacylated form globotriaosylsphingosine (Lyso-GL-3) in multiple organs, causing neural, renal, cardiac, dermatological, gastrointestinal and ophthalmic manifestations, even leading to life-threatening complications. Cardiovascular and cerebrovascular complications (i.e. heart failure, stroke, etc.) or end-stage renal disease even premature death can be seen in severe cases. The life expectancy of male patients is reduced by 15~20 years, while that of female patients is reduced by 6~10 years.

The exact prevalence of FD is currently unknown. Based on an estimated prevalence of 1:60,000, there are approximately 23,000 affected FD patients in China. The clinical manifestations of FD are diverse and non-specific, which may lead to misdiagnosis in patients with non-typical clinical manifestations in the absence of a family history of FD. Cardiac involvement can be recognized in up to 68% patients with FD, significantly higher than in other organs, and the positive screening rate for FD in adults with unexplained left ventricular hypertrophy (LVH)/hypertrophic cardiomyopathy was 0.9%.

Cardiovascular disease is the leading cause of death in patients with FD cardiomyopathy (40.2%). The 2020 Expert Consensus Document on the Management of Cardiovascular Manifestations of Fabry Disease recommends early screening in patients with suspected LVH for early diagnosis. Therefore, strengthened screening strategy in high-risk patients with LVH will improve the diagnosis and treatment of FD in China.

ELIGIBILITY:
Inclusion Criteria:

Patients to be enrolled in this study should fulfill all 3 criteria (a, b, and c) at screening:

1. Patients with a maximum myocardial wall thickness (left ventricular posterior wall or septum) of ≥13 mm at the end diastole on echocardiography;
2. At least two or more "warning signs" associated with FD ("warning signs" include cardiac "warning signs", extracardiac "warning signs", or family history)
3. Aged 18 years old or older;

cardiac "warning signs" of FD:

Concentric LVH or papillary hypertrophy or right ventricular hypertrophy on echocardiography

ECG abnormalities (eg, shortened PR interval, wide QRS complex, right bundle branch block, ST-segment depression, etc.)

Extra-cardiac "warning signs" of FD

Angiokeratomas

Acroparesthesia

Hypohidrosis

Premature stroke (<50 years of age)

Corneal verticillate

Renal impairment accompanied by proteinuria

Hearing loss

Family history

Family history of X-linked inherited disorder (renal disease or cardiac disease)

Exclusion Criteria:

1. LVH patients with a clear etiology;
2. Combining any other clinical condition with a life expectancy less than 1 year;
3. Refuse to give informed consent or refuse to be followed-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a maximum myocardial wall thickness (left ventricular posterior wall or septum) of ≥13 mm at the end diastole on echocardiography, with at least two or more "warning signs" associated with FD ("warning signs" include cardiac "warning signs", extracardiac "warning signs", or family history) who fullfil the standard of screening for Fabry disease will be consecutively recruited.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular deaths | 12 months
  Including sudden cardiac death or equivalent events, heart failure-related death, stroke-related death and death from other cardiovascular causes.

SECONDARY OUTCOMES:
Heart failure | 12 months
  NYHA progression to level III/IV
Stroke | 12 months
  Including ischemic stroke and hemorrhagic stroke
Myocardial infarction | 12 months
  Including ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction
All-cause deaths | 12 months
  Death from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Lei Song, Principal Investigator — Fuwai Hospital, National Centre for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Centre for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No